CLINICAL TRIAL: NCT06874556
Title: Community Paramedic Heart Failure Management (CP-HF) Program
Brief Title: A Study of Paramedic HF Management
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Sara B. Severson, Principal Investigator, Mayo Clinic
Other Study IDs: 24-009568
Record Dates: First submitted 2025-03-03; First posted 2025-03-13 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Community Paramedic Heart Failure Management (CP-HF) program
  Interventions: Behavioral: CP-HF Management
- Standard of Care (SOC)

INTERVENTIONS:
Behavioral: CP-HF Management — Community Paramedics will visit patients up to twice daily. Visits will include patient care discussion with Heart Failure APP, IV placement, lab phlebotomy, heart failure education, and IV medication administration. Community Paramedics will administer up to 120 mg IV furosemide twice daily.
  Groups: Community Paramedic Heart Failure Management (CP-HF) program

SUMMARY:
The purpose of this research is to see if having community paramedic (CP) visit patients at home to manage their heart failure help them stay out of the hospital and improve their overall health compared to standard care. The investigators want to find out if their approach is better for patients in terms of their quality of life, hospital stays, emergency visits, and cost. The investigators are also looking to see how happy patients and doctors are with this method and if it's a practical and sustainable option for the future.

ELIGIBILITY:
Inclusion Criteria:

One of the following criteria:

1. Adults admitted to the hospital with decompensated HF eligible for early discharge with CP support and monitoring.
2. Acutely decompensated HF patients at home or being evaluated in the ambulatory clinic who require large volume diuresis but do not require hospital-level monitoring.
3. Stage D advanced HF patients who require frequent (>weekly) diuretic adjustments (either inpatient or outpatients).

Exclusion Criteria:

1. Hospital-level monitoring or care is clinically indicated.
2. Failed safety assessment, active substance abuse, or behavioral health diagnosis which could impact participation.
3. Enrolled in hospice.
4. Patient is a resident in a skilled nursing facility.
5. Patient does not have a primary care physician or cardiologist at Mayo Clinic.
6. Patient participants with communication barriers due to medical illness or cognitive impairment.
7. Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be identified by the inpatient cardiology services along with outpatient cardiology and/or primary care offices.
Sampling Method: Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2025-06-24 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Number of Days without Hospitalization | From date of randomization until the date of first documented progression or date of death from any cause, whichever comes first, assessed up to 12 months
  Number of Days without Hospitalization will be measured by the number of days a patient is not admitted to the hospital.
Number of Days in the Hospital | From date of randomization until the date of first documented progression or date of death from any cause, whichever comes first, assessed up to 12 months
  Number of Days in the Hospital will be determined by a patient's length of hospital stay.
Number of Emergency Department (ED) Visits | From date of randomization until the date of first documented progression or date of death from any cause, whichever comes first, assessed up to 12 months
  Number of Emergency Department (ED) Visits will be determined by the number of ED visits per patient
Number of Hospitalizations | From date of randomization until the date of first documented progression or date of death from any cause, whichever comes first, assessed up to 12 months
  Number of Hospitalizations will be determined by the number of patients that are hospitalized.
Minnesota Living with Heart Failure Questionnaire (MLHFQ) | Baseline, 31 Days
  Minnesota Living with Heart Failure Questionnaire (MLHFQ) is a 21-question quality of life questionnaire. The scores can range from 0-105, with a higher score reflecting a worse quality of life
Number of patients to comply with the guideline-directed medical therapy (GDMT) | From date of randomization until the date of first documented progression or date of death from any cause, whichever comes first, assessed up to 12 months
  Number of patients to comply with the guideline-directed medical therapy (GDMT) will be measured through medical record reviews to determine changes in adherence rates to prescribed HF medications and therapies.

SECONDARY OUTCOMES:
Patient Satisfaction | up to 1 year
  Measured through a structured patient satisfaction survey developed for the CP-HF program. The survey assesses various aspects of patient experience, including communication, responsiveness, medication management, and overall satisfaction. Responses are rated on a 5-point Likert scale (1 = Strongly Disagree, 5 = Strongly Agree), with higher scores indicating greater satisfaction. Additional questions evaluate care coordination, interpreter service utilization, perceived safety, and willingness to recommend the program.
Clinician Satisfaction | up to 1 year
  Measured through the Clinician & Stakeholder Satisfaction Survey, which assesses clinician experiences and perceptions of the CP-HF program's effectiveness. The survey includes questions on program structure, implementation, sustainability, and collaboration. Responses are rated on a 5-point Likert scale, with higher scores indicating greater satisfaction.
Stakeholder-Perceived Sustainability | up to 1 year
  Stakeholder-Perceived Sustainability will be measured through interviews and surveys of key stakeholders to gauge their views on the sustainability and scalability of the CP-HF program.
Cost-effectiveness of Community Paramedic Program | up to 1 year
  Cost-effectiveness will be determined by comparing the measured cost of the community Paramedic Program against the Standard of Care (SOC)

CONTACTS AND LOCATIONS:
Overall Officials: Sara Severson, APRN, C.N.P., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No